CLINICAL TRIAL: NCT01792323
Title: Subcutaneous Insulin Absorption Following Bolus Administrations With an Insulin Pump - Comparison of Bolus Administrations With Different Bolus Durations
Brief Title: Absorption of Insulin Following Subcutaneous Bolus Administration With Different Bolus Durations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Pieber Thomas, MD, MD, Prof. of Medicine, Medical University of Graz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CIPHER-Clamp
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Type 1 Diabetes
Keywords: insulin pump therapy; insulin bolus; rapid acting insulin; insulin lispro; pharmacodynamics; pharmacokinetics; glucose clamp
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 bolus of insulin lispro with short bolus duration (Experimental): Subcutaneous administration of insulin lispro as a bolus of 15 IU over a period of 30 seconds
  Interventions: Drug: Insulin LISPRO
- 1 bolus of insulin lispro with long bolus duration (Experimental): Subcutaneous administration of insulin lispro as a bolus of 15 IU over a period of 10 minutes
  Interventions: Drug: Insulin LISPRO

INTERVENTIONS:
Drug: Insulin LISPRO — Administration of 15 IU of insulin lispro over a period of 30 seconds

SUMMARY:
To cover meal-related insulin requirements, insulin pumps allow insulin to be delivered at high rates over a short period of time (bolus delivery). The length of this period (bolus duration) usually depends on the chosen bolus size and on the used insulin pump model. This study will evaluate the impact of different bolus durations (i.e., durations commonly employed in commercially available insulin pumps: 2 and 40 seconds for delivering 1 Unit of insulin) on the pharmacokinetic and pharmacodynamic properties of an rapid-acting insulin analogue.

Objective: To evaluate in type 1 diabetic patients the pharmacodynamics and pharmacokinetics of rapid-acting insulin (insulin lispro) administered as subcutaneous boluses with different bolus durations.

Study design: Single-center, randomized, controlled, two-arm cross-over intervention study

Population: Twenty type 1 diabetic subjects

Intervention: The investigational treatment is the subcutaneous administration of insulin lispro either as one bolus of 15 IU over a period of 30s or as one bolus of 15 IU over a period of 10 min. Plasma samples to assess pharmacodynamic and pharmacokinetic properties will be taken during an 8-hour clamp experiment. Patients will undergo both investigational treatments in a randomized order; between the two clamp visits there will be a wash-out period of 5-21 days.

Main study endpoint: Time to maximum glucose infusion rate

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged 18-60 years (both inclusive)
* Type 1 diabetes treated with multiple daily insulin injection or continuous subcutaneous insulin infusion for 12 months
* Fasting C-peptide < 0.3nmol/L
* Body mass index 20.0-30.0 kg/m² (both inclusive)
* HbA1c < 10%

Exclusion Criteria:

* Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods
* Skin pathology or condition prohibiting needle insertion/insulin administration as judged by the investigator
* History of bleeding disorder
* Current participation in another clinical study
* Use of insulin lispro >2 weeks
* Significant acute or chronic illness that might interfere with subject safety or integrity of results as judged by the investigator
* Smoker (defined as >5 cigarettes/d)
* Lipodystrophy
* Current treatment with systemic (oral or i.v.) corticosteroids, monoamine oxidase (MAO) inhibitors, non-selective beta-blockers, growth hormone, herbal products or non-routine vitamins. Furthermore, thyroid hormones are not allowed unless the use of these has been stable during the past 3 months
* Significant history of alcoholism or drug abuse or a positive result in urine drug/alcohol screen

Study Day Exclusion Criteria:

* Strenuous exercise within the last 24 hours prior to the clamp visit
* Non-fasting (i.e. consumption of food or beverages, other than water, later than 22:00 hours the evening before the visit) except if slight intake of rapidly absorbable carbohydrates has been necessary in order to prevent hypoglycaemia
* Injection of long-acting insulin (e.g. insulin glargine or insulin detemir) later than 12:00 hours (noon), 2 days before the clamp visit
* Injection of NPH insulin or other intermediate-acting insulin products later than 12:00 hours (noon) on the day before the clamp visit
* Injection of any short acting insulin (aspart, lispro, glulisine) or more than 6 IU of human insulin between 22:00 hours and 03:00 hours the night before the clamp visit
* Injection of any insulin later than 03:00 hours the night before the clamp visit
* Infusion of any insulin later than 03:00 hours the night before the clamp visit for subjects using continuous subcutaneous insulin infusion (CSII)
* Positive result of alcohol breath test
* Any medical condition that, in the opinion of the Investigator, could interfere with insulin pharmacokinetics and/or glucose metabolism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
tmax(GIR); time to maximum glucose infusion rate | 8 hours

SECONDARY OUTCOMES:
GIRmax, maximum glucose infusion rate | 8 hours

OTHER OUTCOMES:
tmax(ins), time to maximum observed plasma insulin lispro concentration | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, MD, Principal Investigator — Medical University of Graz, Internal Medicine, Endocrinology and Metabolism
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- See also: Medical University of Graz — http://www.medunigraz.at